CLINICAL TRIAL: NCT04567082
Title: Proteome- and Methylation Profiles in Oropharyngeal Cancer
Acronym: PROMEO
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Sander Danstrup, Associate Professor, M.D., Aalborg University Hospital
Other Study IDs: N-20200024
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer group
  Interventions: Diagnostic Test: Examination of saliva
- Control group
  Interventions: Diagnostic Test: Examination of saliva

INTERVENTIONS:
Diagnostic Test: Examination of saliva — Collection of saliva samples

SUMMARY:
This clinical study aims to evaluate proteome- and methylation profiles in saliva in patients with oropharyngeal cancers

ELIGIBILITY:
Cancer group:

Inclusion Criteria:

* Written informed consent
* Verified oropharyngeal squamous cell carcinoma

Exclusion Criteria:

* Other active cancer
* Uncontrolled comorbidity
* Unable to give informed consent

Control group:

Inclusion Criteria:

* Written informed consent
* Normal ENT examination

Exclusion Criteria:

* Active cancer
* Uncontrolled comorbidity
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancergroup:
  Patients from the Northern Region of Denmark referred to the Department of Otolaryngology - Head and Neck Surgery, Aalborg University Hospital with suspected or verified oropharyngeal cancer. Only patients with verified cancer after diagnostic work-up will be included in the analyses.
  Control group:
  Patients referred to the Department of Otolaryngology - Head and neck surgery, Aalborg University Hospital or a private clinic for Oral- and Maxillofacial surgery in Aalborg.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in proteome and methylation profiles | At diagnosis
  Differences between cancer- and control group

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaihede, Professor, Principal Investigator — Department of Otolaryngology - Head and Neck Surgery, Aalborg University Hospital
Locations (1):
- Department of Otolaryngology - Head and Neck Surgery, Aalborg, Denmark